CLINICAL TRIAL: NCT04696705
Title: The Safety and Efficacy Assessment of Ex-Vivo Expanded Allogeneic γδT Cells Immunotherapy in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma (NHL) and Peripheral T Cell Lymphomas (PTCL)
Brief Title: Allogeneic γδ T Cells Immunotherapy in r/r Non-Hodgkin's Lymphoma (NHL) or Peripheral T Cell Lymphomas (PTCL) Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Beijing GD Initiative Cell Therapy Technology Co., Ltd. (Industry); Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zou Dehui, Assistant Director of lymphoma Diagnosis and Treatment Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020028-EC-3
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Non-Hodgkin's Lymphoma (NHL); Peripheral T Cell Lymphoma (PTCL)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic γδT cell immunotherapy (Experimental): Patients will receive 2 cycles of ex-vivo expanded allogeneic γδT cells treatments, at 14 days' intervals, each cycle has 2 infusions. Ex-vivo expanded γδT cells are transfused to patients in a dosage escalated manner (Dose escalation, 1×107, 3×107, 9×107 per kg of body weight).
  Interventions: Biological: Ex-vivo expanded allogeneic γδT cells

INTERVENTIONS:
Biological: Ex-vivo expanded allogeneic γδT cells — Cells will be extracted from a healthy donor by apheresis, followed by ex-vivo expansion and activation. The ex-vivo expanded γδT cells from donors will be adoptively transfused.

SUMMARY:
This study aims to evaluate the safety, tolerability and efficacy of ex-vivo expanded allogeneic γδT cells obtained from a blood-related donor of patients with relapsed or refractory B cell non-Hodgkin's lymphoma (B-NHL) or peripheral T cell lymphoma (PTCL) expect for γδT lymphoma.

DETAILED DESCRIPTION:
This study is a single-center, non-randomized, open label, no control, prospective clinical trial to evaluate the safety, tolerability and efficacy of ex-vivo expanded allogeneic γδT cells from a blood-related donor of NHL or PTCL patients(except for γδT lymphoma). This study will include the following sequential phases: sign informed consent, γδT cell pre-culture, screening and registration to the trial, apheresis, γδT cell preparation, pre-treatment for lymphodepleting chemotherapy (selectable plan), treatments and follow-ups. The study will evaluate the safety and efficacy of the ex-vivo expanded allogeneic γδT cells in patients with relapsed or refractory non-Hodgkin's lymphoma (NHL) or peripheral T cell lymphoma (PTCL) expect for γδT lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient Inclusion Criteria:

  1. Patients should sign informed consent form voluntarily before the trail and comply with the requirements of this study.
  2. Age≥18 years old, gender unlimited.
  3. Patients whose relatives are willing to donate PBMCs voluntarily.
  4. Patients with relapsed or refractory B cell non-Hodgkin's lymphoma (B-NHL) or peripheral T cell lymphoma (PTCL) expect for γδT lymphoma.
  5. Patients had an evaluable imaging lesion of at least greater than 1.5 cm.
  6. Eastern Cooperative Oncology Group (ECOG) Performance score≤2.
  7. Adequate bone marrow function:

     * Absolute neutrophil count (ANC) >1000/mm3;
     * Absolute lymphocyte count (ALC)≥300/mm3;
     * PLT≥50,000/mm3;
     * Hb >8.0g/dl.
  8. Adequate organ function:

     * Alanine aminotransferase (ALT)≤3 times the upper limit of normal (ULN);
     * Aspartate aminotransferase (AST)≤3 times ULN
     * TBIL≤1.5 times ULN (Gilbert syndrome patients TBIL≤3 times ULN and DBIL≤1.5 times ULN)
     * Scr≤1.5 times ULN or CCR≥60 mL/min/1.73m3 Note: apart from tumor infiltrated liver dysfunction.
  9. Male and female patients of reproductive potential must agree to use birth control during the study and for at least 12 weeks post study.
* Donor Inclusion Criteria:

  1. Sign informed consent form.
  2. Age 18 years up to the age of 60 (≤60), gender unlimited.
  3. Relatives of patients (unrestricted to blood relationship).
  4. Apheresis available.
  5. PLT≥100×109/L with normal APTT or PT.

Exclusion Criteria:

* Patient Exclusion Criteria:

  1. Patients with other available treatment drugs or treatment options.
  2. Patients with history of allogeneic hematopoietic stem cell transplantation (Allo-HSCT).
  3. Active central nervous system (CNS) lymphoma.
  4. Patients receiving chemotherapy within 1 week prior to γδT cell transfusion, with the following exceptions:

     * Pretreatment chemotherapy prescribed by the protocol
     * Other exploratory combined medications
  5. Systemic glucocorticoid treatment 72h prior to γδT cell transfusion (apart from physiological replacement dosage).
  6. Biphosphonates were used 2 months prior to γδT cell transfusion.
  7. Patients with systemic vasculitis, or with active or uncontrolled autoimmune diseases, as well as primary or secondary immunodeficiency diseases.
  8. Active HBV, HCV, HIV, TP, CMV or EBV infection.
  9. Major surgery that was evaluated by the investigator as unsuitable for inclusion within 4 weeks prior to screening.
  10. Patients with malignant tumors, apart from those who has been cured for at least 2 years.
  11. Patient's cardiac function meets any of the following conditions:

      * Left ventricular ejection fraction (LVEF)≤45%
      * Class III or IV heart failure according to the NYHA Heart Failure Classifications
      * QTcB>450 msec
      * Other cardiac disease that investigators judge is not suitable for enrollment
  12. History of epilepsy or other active central nervous system disorders.
  13. Inoculated live vaccine within 6 weeks before screening.
  14. Uncontrolled serious active infection (such as sepsis, bacteremia and fungemia).
  15. Life expectancy < 3 months
  16. Participated in any other interventional clinical trial within 3 months prior to γδT cell transfusion.
  17. Any situation that investigators believe the risk of the subjects is increased or results of the trial are disturbed: patients with any serious acute or chronic physical or mental illness, or laboratory abnormalities.
* Donor Exclusion Criteria:

  1. History of any severe clinical diseases or other severe organic diseases, including any history of clinically significant systematic diseases such as cardiovascular, urinary, circulatory, respiratory, neurological, psychiatric, digestive and endocrine diseases. History of high blood pressure or systolic pressure>140 mmHg, diastolic pressure>90 mmHg in screening stage. Any situation that investigators believe is clinically significant or with other severe diseases unsuitable of apheresis.
  2. Arterial thrombosis or venous thrombosis history 12 months prior to the trial or hemorrhagic tendency or history 2 months prior to the trial; oral administration of anticoagulation drugs (e. g. aspirin and warfarin).
  3. Active or history of autoimmune diseases including but not restricted to SLE, psoriasis, RA, IBD and HT. Apart from hypothyrosis which can be controlled by hormone replacement therapy, skin diseases without systemic therapy and celiac disease which is fully controlled.
  4. HIV-Ab, TP-Ab, HCV-Ab, HBsAg, HBeAg, HBeAb or HBcAb positive.
  5. Any symptom, sign or laboratory examination abnormality suggesting acute or subacute infection (e.g. fever, cough, urinary irritation, skin infectious wound).
  6. Female who are pregnant or cannot stop lactating.
  7. Those who cannot communicate with medical staff due to mental illness or language disabilities.
  8. Other unsuitable conditions that investigators believe unsuitable for the donation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2021-12-25 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation: Incidence of Adverse events (AEs) | 2 years post γδT cells infusion
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
Safety evaluation: Dose limited toxicity (DLTs) | 28 days
  The incidence of DLTs will be recorded and assessed.
Safety evaluation: Maximum-tolerated dose (MTD) | 28 days
  MTD or clinical recommended dose will be recorded and evaluated.

SECONDARY OUTCOMES:
Efficacy evaluation：Overall response rate (ORR) | 2 years post γδT cells infusion
  ORR is defined as the incidence of either a CR or a partial response (PR) per the Lugano Classification as determined by study investigators.
Efficacy evaluation：Disease control rate (DCR) | 2 years post γδT cells infusion
  DCR is defined as the incidence of either a CR, a partial response (PR) or stable disease (SD) per the Lugano Classification as determined by study investigators.
Efficacy evaluation：Duration of remission (DOR) | 2 years post γδT cells infusion
  DOR is defined only for participants who experience an objective response after γδT cells infusion and is the time from the first objective response to disease progression or death from any cause.
Efficacy evaluation：Progression free survival (PFS) | 2 years post γδT cells infusion
  PFS is defined as the time from the γδT cells infusion date to the date of disease progression or death from any cause.
Efficacy evaluation：Overall survival (OS) | 2 years post γδT cells infusion
  OS is defined as the time from γδT cells infusion to the date of death from any cause.
Pharmacokinetics (PK) evaluation :γδT cells in peripheral blood | 2 years post γδT cells infusion
  Number of γδT cells in peripheral blood will be assessed by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Zhang, PhD, Study Director — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No